CLINICAL TRIAL: NCT05119530
Title: U.S. POC Study to Evaluate the Performance of the AcuVid COVID-19 Rapid Antigen Saliva Test
Brief Title: POC Study to Evaluate the Performance of the AcuVid COVID-19 Rapid Antigen Saliva Test
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Therma Bright Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: TB20-03
Record Dates: First submitted 2021-11-11; First posted 2021-11-15 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: AcuVid COVID-19 Rapid Antigen Saliva Test — The AcuVid COVID-19 Rapid Antigen Saliva Test is a lateral flow immunoassay to detect SARS-CoV-2 nucleocapsid antigens in human saliva specimens

SUMMARY:
The AcuVid COVID-19 Rapid Antigen Saliva Test is a lateral flow immunoassay to detect SARS-CoV-2 nucleocapsid antigens in human saliva specimens from individuals suspected of COVID-19 by their healthcare provider within the first seven days of symptom onset, or from individuals without symptoms or other epidemiological reasons to suspect.

The AcuVid COVID-19 Rapid Antigen Saliva Test performance will be compared to a high sensitivity FDA EUA approved RT-PCR COVID-19 test. Nasopharyngeal (for RT-PCR) swab results will be collected from subjects by healthcare providers at CLIA Waived COVID-19 Testing Centers, and on the same day the subjects will also provide saliva samples which will be tested and interpreted by the healthcare providers.

This prospective, observational, study will test up to 300 participants to establish the performance characteristics of the AcuVid test on saliva specimens.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing to sign verbal informed consent form.
* Age ≥12 and parents or legal guardians must consent as required by law.
* Participant is attending COVID-19 testing centre to provide a nasopharyngeal swab sample.
* Participant is willing to provide a self-collected saliva sample.

Exclusion Criteria:

* Participant has previously tested positive for COVID-19 within the past 90 days.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will come from individuals visiting COVID-19 testing Centers for the purpose of obtaining a COVID-19 RT-PCR test results. Individuals will be approached to determine eligibility and obtain consent after they have provided a NP swab sample for their COVID-19 RT-PCR test.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Establish performance of AcuVid COVID-19 Rapid Antigen Saliva Test | 1 day
  To establish the performance characteristics of the AcuVid COVID-19 Rapid Antigen Saliva Test in a point-of-care (POC) CLIA Waived setting with lay users (no laboratory experience) testing a participant that has self-collected a saliva specimen. Clinical accuracy of the AcuVid Test will be compared to RT-PCR test results. Accuracy refers to the (PPA, positive percent agreement (sensitivity) and (NPA, negative percent agreement (specificity) between the results of the AcuVid Test and the comparator RT-PCR test.

CONTACTS AND LOCATIONS:
Locations (1):
- Covid Clinic Inc., Modesto, California, United States

IPD SHARING:
Plan to Share IPD: No